CLINICAL TRIAL: NCT02390908
Title: Improving HIV and Alcohol-Related Outcomes Among HIV+ Persons in Clinic Settings
Acronym: PLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Tyrel Starks, Associate Professor, Hunter College of City University of New York
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AA022302 (NIH); R01AA022302 (NIH)
Record Dates: First submitted 2015-03-06; First posted 2015-03-18 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: HIV; Alcohol Use; Medication Adherence
Keywords: alcohol use; hazardous drinking; behavioral intervention; ART adherence; viral load; CD4
MeSH Terms: conditions — Alcohol Drinking; Medication Adherence | interventions — Methods; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Site 1 Immediate PLUS intervention (Experimental): Site 1 Immediate delivery of the PLUS intervention (Six sessions of Motivational Interviewing and Cognitive Behavioral Skills Training)
  Interventions: Behavioral: Immediate PLUS intervention
- Wait-list PLUS condition (Active Comparator): Received the PLUS intervention at 12 months post baseline
  Interventions: Behavioral: Wait-list PLUS intervention
- Site 2 Immediate PLUS intervention (Experimental): Site 2 Immediate delivery of the PLUS intervention (Six sessions of Motivational Interviewing and Cognitive Behavioral Skills Training)
  Interventions: Behavioral: Immediate PLUS intervention
- Site 3 Immediate PLUS intervention (Experimental): Site 3 Immediate delivery of the PLUS intervention (Six sessions of Motivational Interviewing and Cognitive Behavioral Skills Training)
  Interventions: Behavioral: Immediate PLUS intervention

INTERVENTIONS:
Behavioral: Immediate PLUS intervention — The Positive Living through Understanding and Support (PLUS) intervention consists of six sessions that utilizes motivational interviewing and cognitive behavioral skills training to reduce alcohol use and improve medication adherence.
  Arms: Site 1 Immediate PLUS intervention; Site 2 Immediate PLUS intervention; Site 3 Immediate PLUS intervention
Behavioral: Wait-list PLUS intervention — In addition to treatment as usual, participants will receive handouts with printed information about HIV, the importance of ART adherence, and problematic alcohol use and HIV disease progression. Following their assessment 12 months after their baseline visit, participants will receive the PLUS intervention.
  Arms: Wait-list PLUS condition

SUMMARY:
Alcohol use is increasingly recognized as a key factor in morbidity and mortality among HIV-positive individuals and represents an important public health concern, given its associations with medication non-adherence, increases in viral load, poor immunologic outcomes (lower cluster of differentiation 4, or CD4, counts), drug resistance, lower health care utilization, comorbidities (HIV/viral hepatitis coinfection), and poor health outcomes overall. Adherence to HIV medications has a double public health benefit, both in terms of slowing disease progression and improving health outcomes among HIV-positive individuals and in helping to curb the sexual transmission of HIV. The objective of this study is to implement a multisite comparative effectiveness trial in real-world clinical settings with three intensities of treatment to test the clinical and cost effectiveness of an efficacious, theory-based behavioral intervention (PLUS) in improving adherence to antiretroviral therapy (ART) and alcohol-related outcomes among HIV-positive individuals who drink alcohol at harmful or hazardous levels. The study is being conducted in collaboration between the Center for HIV Educational Studies and Training (CHEST) at Hunter College at the City University of New York (CUNY) and the Spencer Cox Center for Health at the Institute for Advanced Medicine, Mount Sinai Health System.

DETAILED DESCRIPTION:
Alcohol consumption at harmful or hazardous levels among HIV-positive persons exacerbates health problems and accelerates HIV disease progression. Antiretroviral therapy (ART) has been the single most important treatment for people living with HIV to optimize viral suppression and slow disease progression. Adherence to ART has considerable public health implications, particularly given that optimal adherence decreases morbidity and mortality, decreases the potential for the development of drug resistant strains of HIV, and reduces HIV infectiousness.

Project PLUS (Positive Living through Understanding and Support) was the first (and to our knowledge only) theory-based behavioral intervention, which integrates motivational interviewing and cognitive-behavioral skills training, to demonstrate significant improvements in viral load, CD4 cell count, and self-reported adherence among a racially and ethnically diverse sample of HIV-positive women and men enrolled in a randomized controlled trial, and the first intervention for hazardous drinkers to demonstrate any significant effects. A clinic-based replication is the crucial next step in studying the intervention's effectiveness in the real world when delivered by HIV clinic providers to their patients.

In collaboration with medical providers at the Spencer Cox Center for Health at the Institute for Advanced Medicine, Mount Sinai Health System, the largest provider of HIV medical care in the New York City area, our goals are to better understand alcohol-related outcomes among HIV-positive persons over the lifespan and to conduct a multisite comparative effectiveness trial with three intensities of treatment-the PLUS intervention, an enhanced treatment as usual (eTAU) condition, and treatment as usual (TAU) condition-to test the clinical and cost-effectiveness of the PLUS intervention in reducing alcohol use and improving ART adherence, viral load, and CD4 counts among HIV-positive hazardous drinkers. This study has the potential to exert a sustained and powerful impact on the effectiveness of ART interventions for HIV-positive persons with problematic drinking.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Currently receiving ART
* Current viral load (VL) ˃200 copies/ml
* Report drinking at hazardous levels, operationalized as exceeding 14 standard drinks per week for men or exceeding 7 standard drinks per week for women, or reported use of illicit drugs exclusive of marijuana or illicit use of prescription opioids within the past 3 months.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyrel J Starks, PhD, Principal Investigator — Hunter College of City University of New York
Locations (1):
- Center for HIV/AIDS Educational Studies and Training of Hunter College, CUNY, New York, New York, United States

REFERENCES:
- [Background] Parsons JT, Golub SA, Rosof E, Holder C. Motivational interviewing and cognitive-behavioral intervention to improve HIV medication adherence among hazardous drinkers: a randomized controlled trial. J Acquir Immune Defic Syndr. 2007 Dec 1;46(4):443-50. doi: 10.1097/qai.0b013e318158a461. PMID 18077833
- [Derived] Starks TJ, Skeen SJ, Scott Jones S, Gurung S, Millar BM, Ferraris C, Ventuneac A, Parsons JT, Sparks MA. Effectiveness of a Combined Motivational Interviewing and Cognitive Behavioral Intervention to Reduce Substance Use and Improve HIV-Related Immune Functioning. AIDS Behav. 2022 Apr;26(4):1138-1152. doi: 10.1007/s10461-021-03467-7. Epub 2021 Sep 19. PMID 34537912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 174 participants were enrolled in the experimental arms of PLUS. An additional 120 comparison patients, in regular care at sites but not enrolled in the study, had their electronic medical records (EMR) accessed. They were not considered enrolled in the study, as they did not sign informed consent, and did not receive intervention. Data for this "No-Treatment EMR Control" group included viral load, CD4 and demographics but not study measures (alcohol and drug use severity, medication adherence).
Groups:
- Site 1 Immediate PLUS Intervention; Site 2 Immediate PLUS Intervention; Site 3 Immediate PLUS Intervention: Immediate delivery of the PLUS intervention (Six sessions of Motivational Interviewing and Cognitive Behavioral Skills Training)
  Immediate PLUS intervention: The Positive Living through Understanding and Support (PLUS) intervention consists of six sessions that utilizes motivational interviewing and cognitive behavioral skills training to reduce alcohol use and improve medication adherence.
- Wait-list PLUS Condition: Received the PLUS intervention at 12 months post-baseline
  PLUS intervention: The Positive Living through Understanding and Support (PLUS) intervention consists of six sessions that utilizes motivational interviewing and cognitive behavioral skills training to reduce alcohol use and improve medication adherence.
  Wait-list PLUS intervention: In addition to treatment as usual, participants will receive handouts with printed information about HIV, the importance of ART adherence, and problematic alcohol use and HIV disease progression. Following their assessment 12 months after their baseline visit, participants will receive the PLUS intervention.
- No-Treatment EMR Control Group: The EMRs of randomly selected patients who belonged to the TAU site and were not enrolled in the PLUS trial were matched on key patient characteristics for comparisons with EMRs of patients in the PLUS intervention and Waitlist control conditions. This matched cohort of patients received care at a fourth clinic that did not receive any intervention (i.e., PLUS or eTAU) and was considered as a natural history comparison group.
  This group were only included in analyses comparing VL and CD4.
Period: Overall Study
Arm/Group | Site 1 Immediate PLUS Intervention | Site 2 Immediate PLUS Intervention | Site 3 Immediate PLUS Intervention | Wait-list PLUS Condition | No-Treatment EMR Control Group
Started | 40 | 22 | 22 | 90 | 120
Completed | 40 | 22 | 22 | 90 | 120
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Wait-list PLUS Condition: Received the PLUS intervention at 12 months post baseline
  PLUS intervention: The Positive Living through Understanding and Support (PLUS) intervention consists of six sessions that utilizes motivational interviewing and cognitive behavioral skills training to reduce alcohol use and improve medication adherence.
  Wait-list PLUS intervention: In addition to treatment as usual, participants will receive handouts with printed information about HIV, the importance of ART adherence, and problematic alcohol use and HIV disease progression. Following their assessment 12 months after their baseline visit, participants will receive the PLUS intervention.
- No-Treatment EMR Control Group: Patients whose electronic medical records (EMRs) were extracted for viral load and CD4 outcomes over the study period, but who were not enrolled in PLUS and did not receive the intervention.
- Total: Total of all reporting groups
Arm/Group | Site 1 Immediate PLUS Intervention | Site 2 Immediate PLUS Intervention | Site 3 Immediate PLUS Intervention | Wait-list PLUS Condition | No-Treatment EMR Control Group | Total
Number analyzed (Participants) | 40 | 22 | 22 | 90 | 120 | 294
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 21 | 22 | 87 | 119 | 288
  >=65 years | 1 | 1 | 0 | 3 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (11.5) | 41.2 (11.3) | 44.0 (10.2) | 45.5 (11.9) | 45.2 (10.7) | 44.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 8 | 20 | 21 | 54
  Male | 38 | 19 | 14 | 70 | 99 | 240
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 18 | 10 | 15 | 51 | 62 | 156
  Race/Ethnicity: Latino | 8 | 8 | 3 | 22 | 21 | 62
  Race/Ethnicity: Other | 7 | 4 | 1 | 9 | 21 | 42
  Race/Ethnicity: White | 7 | 0 | 3 | 8 | 16 | 34
Region of Enrollment [Number; unit: participants]
  United States | 40 | 22 | 22 | 90 | 120 | 174
Drug Use DAST Score [Mean (Standard Deviation); unit: units on a scale] — Drug Abuse Screening Test (DAST-10; Skinner, 1982). This measure was used to characterize a participant's drug use and consequences in the past three months. Participants respond yes (yes = 1) or no (no = 0) to nine items such as "Are you always able to stop using drugs when you want to?". Total/summed scores on the DAST-10 range from 0 to 9, with higher scores indicating greater drug use and associated problems. Population: Drug Use data is only available for the 174 participants who received the intervention. The 120 patients whose EMR records were extracted for viral load and CD4 results did not have data for this variable and were thus not included in analyses.
  units on a scale
    number analyzed (Participants) | 40 | 22 | 22 | 90 | 0 | 174
    (all) | 4.1 (2.7) | 4.0 (2.5) | 2.8 (2.3) | 3.74 (2.7) |  | 3.74 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Viral Load
Description: Standard of care HIV-1 viral load results were run using local laboratories and results were abstracted from EMR data, indicating the participant's most recent viral load result. Each viral load result indicates the number of HIV copies in a milliliter (copies/mL), and raw values were log-transformed to deal with non-normal distribution. Minimum and maximum log-viral load values in the current sample were 1.28 and 6.07, respectively.
Time Frame: most recent result within past 90 days
Measure: Mean (Standard Deviation); unit: Log-transformed copies per. milimeter
Groups:
- No-Treatment Control EMR Group: 120 matched patients in the No-Treatment Control Group whose Viral Load results were obtained through Electronic Medical Records (EMR)
Arm/Group | Site 1 Immediate PLUS Intervention | Site 2 Immediate PLUS Intervention | Site 3 Immediate PLUS Intervention | Wait-list PLUS Condition | No-Treatment Control EMR Group
Number analyzed (Participants) | 40 | 22 | 22 | 90 | 120
Log-transformed copies per. milimeter | 3.1 (1.7) | 1.8 (1.0) | 1.8 (0.6) | 2.6 (1.4) | 2.5 (1.4)
Statistical Analysis 1: Comparison: Site 1 Immediate PLUS Intervention vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.39, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The intercept quoted here represents the difference between Site 1 and the No-Treatment Group at the 3-month follow-up; Analysis adjusted for gender and pre-baseline value of the outcome; Beta = 0.22, 95% CI 2-sided [-0.28 to 0.72] — The main effect of receiving the PLUS intervention at Site 1 on log-transformed Viral Load was estimated against the No-Treatment Control EMR Group
Statistical Analysis 2: Comparison: Site 2 Immediate PLUS Intervention vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.94, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The intercept quoted here represents the difference between Site 2 and the No-Treatment Group at the 3-month follow-up; Analysis adjusted for gender and pre-baseline value of the outcome; Beta = -0.03, 95% CI 2-sided [-0.84 to 0.79] — The main effect of receiving the PLUS intervention at Site 2 on log-transformed Viral Load was estimated against the No-Treatment Control EMR Group
Statistical Analysis 3: Comparison: Site 3 Immediate PLUS Intervention vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.95, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The intercept quoted here represents the difference between Site 3's Immediate Delivery Group and the No-Treatment Group at the 3-month follow-up; Analysis adjusted for gender and pre-baseline value of the outcome; Beta = 0.02, 95% CI 2-sided [-0.69 to 0.74] — The main effect of receiving the PLUS intervention at Site 3 on log-transformed Viral Load was estimated against the No-Treatment Control EMR Group
Statistical Analysis 4: Comparison: Wait-list PLUS Condition vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.09, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The intercept quoted here represents the difference between Site 3 (the Waitlist condition) and the No-Treatment Group at the 3-month follow-up; Analysis adjusted for gender and pre-baseline value of the outcome; Beta = -0.32, 95% CI 2-sided [-0.69 to 0.05] — The main effect of being in the Waitlist condition (i.e., not receiving the PLUS intervention at Site 3) on log-transformed Viral Load was estimated against the No-Treatment Control EMR Group
Statistical Analysis 5: Comparison: Site 1 Immediate PLUS Intervention vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.79, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 1 estimated here represents linear change in log VL across the 3-,6-,9- and 12-month follow-ups for Site 1 relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = -0.03, 95% CI 2-sided [-0.24 to 0.18]
Statistical Analysis 6: Comparison: Site 2 Immediate PLUS Intervention vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.57, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 1 estimated here represents linear change in log VL across the 3-,6-,9- and 12-month follow-ups for Site 2 relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = -0.12, 95% CI 2-sided [-0.53 to 0.36]
Statistical Analysis 7: Comparison: Site 3 Immediate PLUS Intervention vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.97, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 1 here represents linear change in log VL across the 3-,6-,9- and 12-month follow-ups for Site 3 (Immediate) relative to the No-Treatment EMR Control; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = 0.01, 95% CI 2-sided [-0.35 to 0.36]
Statistical Analysis 8: Comparison: Wait-list PLUS Condition vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.41, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 1 estimated here represents linear change in log VL across the 3-,6-,9- and 12-month follow-ups for Waitlist relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = 0.07, 95% CI 2-sided [-0.10 to 0.24]
Statistical Analysis 9: Comparison: Site 1 Immediate PLUS Intervention vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.82, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 2 estimated here represents linear change in log VL across the 12-,15-, and 18-month follow-ups for Site 1 relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = 0.06, 95% CI 2-sided [-0.41 to 0.52]
Statistical Analysis 10: Comparison: Site 2 Immediate PLUS Intervention vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.49, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 2 estimated here represents linear change in log VL across the 12-,15-, and 18-month follow-ups for Site 2 relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = 0.14, 95% CI 2-sided [-0.26 to 0.53]
Statistical Analysis 11: Comparison: Site 3 Immediate PLUS Intervention vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.18, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 2 estimated here represents linear change in log VL across the 12-,15-, and 18-month follow-ups for Site 3 relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = -0.33, 95% CI 2-sided [-0.80 to 0.15]
Statistical Analysis 12: Comparison: Wait-list PLUS Condition vs No-Treatment Control EMR Group; Test type: Superiority; p = 0.89, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 2 estimated here represents linear change in log VL across the 12-,15-, and 18-month follow-ups for Waitlist relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = 0.02, 95% CI 2-sided [-0.28 to 0.32]

2. Primary Outcome: CD4 Count
Description: CD4 results were accessed through clinic EMR data, and represent cells per cubic millimeter.
Time Frame: most recent result within past 90 days
Measure: Mean (Standard Deviation); unit: number of cells per cubic milimeter
Arm/Group | Site 1 Immediate PLUS Intervention | Site 2 Immediate PLUS Intervention | Site 3 Immediate PLUS Intervention | Wait-list PLUS Condition | No-Treatment EMR Control Group
Number analyzed (Participants) | 40 | 22 | 22 | 90 | 120
number of cells per cubic milimeter | 632.4 (355.1) | 696.2 (356.2) | 390.5 (462.9) | 398.2 (252.2) | 409.1 (254.7)
Statistical Analysis 1: Comparison: Site 1 Immediate PLUS Intervention vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.95, Latent Growth Curve — [p-value comment as in outcome 1, analysis 1]; Analysis adjusted for gender and pre-baseline value of the outcome; Beta = 1.92, 95% CI 2-sided [-54.68 to 58.53] — The main effect of receiving the PLUS intervention at Site 1 on CD4 Count was estimated against the No-Treatment Control EMR Group
Statistical Analysis 2: Comparison: Site 2 Immediate PLUS Intervention vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.61, Latent Growth Curve — [p-value comment as in outcome 1, analysis 2]; Analysis adjusted for gender and pre-baseline value of the outcome; Beta = 23.99, 95% CI 2-sided [-67.54 to 115.51] — The main effect of receiving the PLUS intervention at Site 2 on CD4 Count was estimated against the No-Treatment Control EMR Group
Statistical Analysis 3: Comparison: Site 3 Immediate PLUS Intervention vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.48, Latent Growth Curve — [p-value comment as in outcome 1, analysis 3]; Analysis adjusted for gender and pre-baseline value of the outcome; Beta = -23.71, 95% CI 2-sided [-88.82 to 41.40] — The main effect of receiving the PLUS intervention at Site 3 on CD4 Count was estimated against the No-Treatment Control EMR Group
Statistical Analysis 4: Comparison: Wait-list PLUS Condition vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.88, Latent Growth Curve — [p-value comment as in outcome 1, analysis 4]; Analysis adjusted for gender and pre-baseline value of the outcome; Beta = 4.19, 95% CI 2-sided [-49.76 to 58.14] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Site 1 Immediate PLUS Intervention vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.59, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 1 estimated here represents linear change in CD4 count across the 3-,6-,9- and 12-month follow-ups for Site 1 relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = 7.67, 95% CI 2-sided [-19.88 to 35.21]
Statistical Analysis 6: Comparison: Site 2 Immediate PLUS Intervention vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.24, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 1 estimated here represents linear change in CD4 count across the 3-,6-,9- and 12-month follow-ups for Site 2 relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = -24.95, 95% CI 2-sided [-66.78 to 16.88]
Statistical Analysis 7: Comparison: Site 3 Immediate PLUS Intervention vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.15, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 1 estimated here represents linear change in CD4 count across the 3-,6-,9- and 12-month follow-ups for Site 3 relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = 18.32, 95% CI 2-sided [-6.63 to 43.27]
Statistical Analysis 8: Comparison: Wait-list PLUS Condition vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.33, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 1 estimated here represents linear change in CD4 count across the 3-,6-,9- and 12-month follow-ups for Waitlist relative to No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = 10.27, 95% CI 2-sided [-10.20 to 30.74]
Statistical Analysis 9: Comparison: Site 1 Immediate PLUS Intervention vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.80, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 2 estimated here represents linear change in CD4 count across the 12-,15-, and 18-month follow-ups for Site 1 relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = 6.42, 95% CI 2-sided [-44.24 to 57.09]
Statistical Analysis 10: Comparison: Site 2 Immediate PLUS Intervention vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.89, Latent Growth Curve — Piecemeal latent growth curves (LGC) were specified with intercepts and linear slopes. Slope 2 estimated here represents linear change in CD4 count across the 12-,15-, and 18-month follow-ups for Site 2 relative to the No-Treatment EMR Control Group; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = -5.43, 95% CI 2-sided [-85.47 to 74.61]
Statistical Analysis 11: Comparison: Site 3 Immediate PLUS Intervention vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.97, Latent Growth Curve — [p-value comment as in outcome 1, analysis 11]; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = 1.16, 95% CI 2-sided [-60.61 to 62.94]
Statistical Analysis 12: Comparison: Wait-list PLUS Condition vs No-Treatment EMR Control Group; Test type: Superiority; p = 0.07, Latent Growth Curve — [p-value comment as in outcome 1, analysis 12]; Analysis adjusted for gender and pre-baseline value of the outcome; Slope = -38.40, 95% CI 2-sided [-79.51 to 2.72]

3. Primary Outcome: ART Medication Adherence
Description: Percentage of antiretroviral medication (ART) doses that were taken as prescribed, within the past 30 days. Minimum and maximum values were 0% and 100%, respectively.
Time Frame: past 30 days
Measure: Mean (Standard Deviation); unit: percentage of adherent days
Arm/Group | Site 1 Immediate PLUS Intervention | Site 2 Immediate PLUS Intervention | Site 3 Immediate PLUS Intervention | Wait-list PLUS Condition
Number analyzed (Participants) | 40 | 22 | 22 | 90
percentage of adherent days | 85.5 (31.1) | 86.6 (15.8) | 83.4 (18.5) | 77.6 (34.0)
Statistical Analysis 1: Comparison: Site 1 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.22, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The intercept quoted here represents the difference between Site 1 and the Waitlist Group at the 3-month follow-up; Analysis adjusted for gender and pre-baseline value of the outcome; Beta = -7.87, 95% CI 2-sided [-20.52 to 4.78] — The main effect of receiving the PLUS intervention at Site 1 on ART Medication Adherence was estimated against Site 3's Waitlist Control Group
Statistical Analysis 2: Comparison: Site 2 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.22, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The intercept quoted here represents the difference between Site 2 and the Waitlist Group at the 3-month follow-up; Analysis adjusted for gender and pre-baseline value of the outcome; Beta = 10.29, 95% CI 2-sided [-6.25 to 26.82] — The main effect of receiving the PLUS intervention at Site 2 on ART Medication Adherence was estimated against Site 3's Waitlist Control Group
Statistical Analysis 3: Comparison: Site 3 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.96, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The intercept quoted here represents the difference between Site 3's Immediate Delivery Group and the Waitlist Group at the 3-month follow-up; Analysis adjusted for gender and baseline value of the outcome; Beta = -0.27, 95% CI 2-sided [-11.63 to 11.08] — The main effect of receiving the PLUS intervention immediately at Site 3 on ART Medication Adherence was estimated against Site 3's Waitlist Control Group
Statistical Analysis 4: Comparison: Site 1 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.03, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The slope estimated here represents linear change in Medication Adherence across the 3-, 6-, 9- and 12-month follow-ups for Site 1 relative to Waitlist Control Group; Analysis adjusted for gender and baseline value of the outcome; Slope = 6.34, 95% CI 2-sided [0.72 to 11.97]
Statistical Analysis 5: Comparison: Site 2 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.42, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The slope estimated here represents linear change in Medication Adherence across the 3-, 6-, 9- and 12-month follow-ups for Site 2 relative to Waitlist Control Group; Analysis adjusted for gender and baseline value of the outcome; Slope = 3.35, 95% CI 2-sided [-4.78 to 11.47]
Statistical Analysis 6: Comparison: Site 3 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.91, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The slope estimated here represents linear change in Medication Adherence across 3-,6-,9- and 12-month follow-ups for Site 3 (Immediate) relative to Waitlist Control Group; Analysis adjusted for gender and baseline value of the outcome; Slope = 0.34, 95% CI 2-sided [-5.85 to 6.54]

4. Primary Outcome: Alcohol Use Severity
Description: Severity of alcohol consumption as measured by the Alcohol Use Disorders Identification Test (AUDIT). The AUDIT is a 10-item, widely-used screening questionnaire consisting of three questions related to drinking frequency, three questions on dependence, and four questions on problems caused by alcohol over the past three months. Scores range from 0 to 40, with higher scores indicating greater alcohol use.
Time Frame: past 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Site 1 Immediate PLUS Intervention | Site 2 Immediate PLUS Intervention | Site 3 Immediate PLUS Intervention | Wait-list PLUS Condition
Number analyzed (Participants) | 40 | 22 | 22 | 90
score on a scale | 10.38 (6.6) | 3.29 (5.5) | 9.05 (9.6) | 5.93 (6.3)
Statistical Analysis 1: Comparison: Site 1 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.02, Latent Growth Curve — [p-value comment as in outcome 3, analysis 1]; Analysis adjusted for gender and baseline value of the outcome; Beta = 3.19, 95% CI 2-sided [0.61 to 5.78] — The main effect of receiving the PLUS intervention at Site 1 on Alcohol Use severity (AUDIT) was estimated against Site 3's Waitlist Control Group
Statistical Analysis 2: Comparison: Site 2 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.63, Latent Growth Curve — [p-value comment as in outcome 3, analysis 2]; Analysis adjusted for gender and baseline value of the outcome; Beta = -0.86, 95% CI 2-sided [-4.33 to 2.61] — The main effect of receiving the PLUS intervention at Site 2 on Alcohol Use severity (AUDIT) was estimated against Site 3's Waitlist Control Group
Statistical Analysis 3: Comparison: Site 3 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.02, Latent Growth Curve — [p-value comment as in outcome 3, analysis 3]; Analysis adjusted for gender and baseline value of the outcome; Beta = 4.17, 95% CI 2-sided [0.80 to 7.54] — The main effect of receiving the PLUS intervention immediately at Site 3 on Alcohol Use severity (AUDIT) was estimated against Site 3's Waitlist Control Group
Statistical Analysis 4: Comparison: Site 1 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.46, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The slope estimated here represents linear change in AUDIT across the 3-, 6-, 9- and 12-month follow-ups for Site 1 relative to that for the Waitlist Control Group; Analysis adjusted for gender and baseline value of the outcome; Slope = -0.40, 95% CI 2-sided [-1.47 to 0.67]
Statistical Analysis 5: Comparison: Site 2 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.50, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The slope estimated here represents linear change in AUDIT across the 3-, 6-, 9- and 12-month follow-ups for Site 2 relative to that for the Waitlist Control Group; Analysis adjusted for gender and baseline value of the outcome; Slope = -0.29, 95% CI 2-sided [-1.12 to 0.55]
Statistical Analysis 6: Comparison: Site 3 Immediate PLUS Intervention vs Wait-list PLUS Condition; Test type: Superiority; p = 0.43, Latent Growth Curve — A latent growth curve (LGC) with an intercept and linear slope was specified. The slope estimated here represents linear change in AUDIT across the 3-, 6-, 9- and 12-month follow-ups for Site 3 (Immediate) relative to Waitlist Control Group; Analysis adjusted for gender and baseline value of the outcome; Slope = -0.35, 95% CI 2-sided [-1.23 to 0.52]

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- No-Treatment EMR Control Group: Patients not enrolled in PLUS and did not receive the intervention, and were not monitored for adverse events (and thus, no data exists in this regard).
Arm/Group | Site 1 Immediate PLUS Intervention | Site 2 Immediate PLUS Intervention | Site 3 Immediate PLUS Intervention | Wait-list PLUS Condition | No-Treatment EMR Control Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/22 | 1/22 | 3/90 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/22 | 0/22 | 0/90 | 0/120
Other Adverse Events (participants affected / at risk) | 0/40 | 0/22 | 0/22 | 0/90 | 0/120

LIMITATIONS AND CAVEATS:
The sample was recruited in a major metropolitan area and may not be representative of the wider HIV-positive US population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT02390908/Prot_SAP_000.pdf